CLINICAL TRIAL: NCT04769882
Title: Use of the Er:YAG Laser in Conservative Dentistry: Evaluation of the Microbial Population in Carious Lesions
Brief Title: Er:YAG Laser Effects on Microbial Population in Conservative Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Guido Lombardo, University Researcher, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COU003
Record Dates: First submitted 2021-02-14; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Dental Caries; Microbial Colonization
Keywords: Er:YAG Laser; Oral Microbiota; Conservative Dentistry
MeSH Terms: conditions — Dental Caries; Communicable Diseases | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned with a software (Excel 2007) to two groups: group A, control group, which includes treatment with traditional therapy; group B, intervention group, which includes treatment with Er:YAG laser therapy.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: To ensure confidentiality of the data, each subject will be assigned a serial number so that only one of the experimenters will be able to link a number to the corresponding person. In addition, a dedicated computer will be used for data collection and analysis, which will be set up to allow limited access with a password known only to one of the experimenters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er:YAG laser therapy group (Active Comparator): The removal of caries was performed with Er:YAG laser (Doctor Smile, Lambda SRL,Italy) with BOOST handpiece to cut the enamel and open the cavity, and 90° handpiece to remove the carious dentin with tips of 800 µ in diameter and 8 mm or 12 mm in length, in relation to the depth and distance of the lesion.
  Interventions: Device: Er:YAG Laser
- Traditional therapy group (No Intervention): The removal of caries was performed with manual and rotating instruments, such as dentin spoon (ASA Dental S.p.a.), turbine (NSK Dental Italy S.r.l.) with diamond burs (Kerr Dental Italia S.r.l.) to cut the enamel and open the cavity and drill handpiece (KaVo Dental Italia S.r.l.) with tungsten carbide burs (Kerr Dental Italia S.r.l.) to remove the infected dentin.

INTERVENTIONS:
Device: Er:YAG Laser — Selected Er:YAG settings: "enamel removal" program for adult, with "normal" modality (frequency: 20 Hz, energy: 400 mJ, power: 8.0 W, air: 80%, water: 60%) and "dentin removal" program for adult, with "normal" modality (frequency: 20 Hz, energy: 200 mJ, power: 4.0 W, air: 90%, water: 30%)
  Arms: Er:YAG laser therapy group

SUMMARY:
The aim of this study is to verify the quantitative and qualitative effect of Erbium dental laser therapy on microbial populations in carious lesions and to compare the laser therapy with traditional conservative therapies.

DETAILED DESCRIPTION:
Patients will be assessed and selected at the University Odontostomatology Clinic (COU) in Perugia; patients are considered eligible for enrolment if they are at least 18 years old and have a carious lesion on permanent teeth, cavitated and non-destructive, deepening to the middle third of the dentine and no further. The patients will be randomly assigned to two groups as follows: group A, control group, which includes treatment with traditional therapy; group B, intervention group, which includes treatment with Er:YAG laser therapy. For each patient, two salivary swabs will be taken on the cavity dentine of the carious lesion: one before and one after the treatments.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients of both sexes with at least 18 years of age and one cavitated non-destructive carious occlusal lesion of a permanent teeth, that deepens up to the middle third of the dentin and not beyond, confirmed by radiographic exam and without pulp involvement.

Exclusion Criteria:

* patients that refused to sign the informed consent document;
* children or individuals with less than 18 years;
* pregnant subjects;
* patients with syndromes or chronic systemic diseases;
* patients who had used antibiotics within the previous three months or under pharmacological treatments;
* patients with painful symptoms consistent with irreversible pulpitis or mobility and destructive carious lesions extending beyond the middle third of the dentin;
* teeth with exposure of the dental pulp or periodontitis;
* patients with caries on deciduous teeth;
* patients with no cooperation during the radiographical exam and/or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Comparison of microbial load change after Er:YAG and conventional treatments | Measuring before any treatment and after treatments, through study completion, an average of 6 months
  Swabbing of two samples from the cavity floor of lesions: before any treatment and after treatments (laser and traditional). Quantitative evaluation of the microbial population, in terms of Colony Forming Unit (CFU) by seeding the swabs taken in various types of media (Chocolate Agar, CNA Agar, Haemophilus Agar, Sabouraud, McConkey Agar, Shaedler Agar) and analysing the changes from baseline CFUs before any treatment and after Er:YAG laser and conventional therapies (control group and intervention group), comparing the effects of the two different types of treatment .
Comparison of the effects of Er:YAG and conventional therapy in modifying the reduction of specific microbial species through mass spectrometry typing | Measuring before any treatment and after treatments, through study completion, an average of 6 months
  Qualitative evaluation of the microbial species grown by mass spectrometry typing (MALDI TOF MS, Biomèrieux) of colonies freshly collected on culture plates, and analysis of the changes from baseline growth before any treatment and after Er:YAG laser and conventional therapies (control group and intervention group), comparing the effects on the growth of specific microbial populations of the two different types of treatment .

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cianetti, Study Director — Department of Medicine and Surgery
Locations (1):
- University Dental Clinic (C.O.U., Centro Odontostomatologico Universitario) of the University of Perugia, Perugia, Italy